CLINICAL TRIAL: NCT05207839
Title: Randomized, Double-blind Trial Evaluating the Impact of the Consumption of GOS (Galacto Oligosacharides) on the Adult Microbiome
Brief Title: Impact of Galacto-Oligosaccharides on Adult Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2106NRC1
Record Dates: First submitted 2021-10-14; First posted 2022-01-26 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Healthy
MeSH Terms: interventions — Refit milk powder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Milk powder without GOS (Placebo Comparator)
  Interventions: Dietary Supplement: Milk powder
- Milk powder with GOS (Active Comparator)
  Interventions: Dietary Supplement: Milk powder

INTERVENTIONS:
Dietary Supplement: Milk powder — one sachet per day dissolved in 200 ml of water

SUMMARY:
The aim of this study is to evaluate the bifidogenic effect and other potentially beneficial effects on the microbiome of GOS.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years,
* Healthy participants, both male and female
* BMI in the normal and overweight range 18.5 ≤ BMI ≤ 29.9 kg/m2
* Able to understand and to sign a written informed consent prior to study enrolment

Exclusion Criteria:

* Known chronic diseases or conditions for which the investigators/investigation team deem as not suitable for study participation,
* Known food allergy and intolerance e.g. lactose intolerance,
* Habitually, have < 5 spontaneous bowel movements on average per week,
* Chronic or recurrent diarrhoea with spontaneous bowel movements > 2 per day
* Prior gastrointestinal surgery (apart from appendectomy or herniotomy),
* Received systemic antiviral/antibacterial/antifungal therapy during the 3 months prior to study enrolment,
* Medications or supplements that are known to alter gut function or microflora i.e. acid antisecretory drugs, pre-/probiotics, laxative during the 4 weeks prior to study enrolment,
* Anti-hyperlipidaemic, antihypertensive medications and/or anticoagulant agents,
* Currently participating in another interventional clinical trial or research project,
* Alcohol intake > 2 servings per day; specifically, a serving is 0.4 dl of strong alcohols, 1 dl of red or white wine, or 3 dl of beer. Or other chronic substance abuse,
* Changing diet patterns due to travelling and staying abroad for more than two weeks (Asia, Africa, or Latin America) during the two months prior to study enrolment,
* Food restrictions such as vegan, vegetarian, ketogenic, low carb, paleo, raw diets, caloric restrictive diets,
* Artificially sweetened beverage intake >1000 ml/ per day,
* Female participants will be excluded if they are pregnant, have given birth in the last 6 months, or are lactating,
* Subject having a hierarchical or family link with the research team members,
* Occurrence of fever episodes, infection, or vaccination during 14 days before the start of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Proportion of Bifidobacteria in the stools | Throughout 14 days of product intake
  Measured by Next Generation Sequencing (NGS)

SECONDARY OUTCOMES:
Change in quality of life using SF-36 questionnaire (Short Form 36 Health Survey) | Throughout 14 days of product intake
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and are now widely utilized by managed care organizations and by Medicare for routine monitoring and assessment of care outcomes in adult patients. Score ranging from 0 to 100 (higher scores indicate better health status).
Change in Short Chain Fatty Acids (SCFA) in the plasma | Throughout 14 days of product intake
  The SFCA are measured in the plasma using Liquid Chromatography with tandem mass spectrometry (LC-MSMS)
Gastrointestinal Symptom Rating Scale (GSRS) | Throughout 14 days of product intake
  Validated questionnaire exploring the presence and severity of GI symptoms over the previous 7 days. The GSRS is a disease-specific instrument of 15 items combined into five symptom clusters depicting reflux, abdominal pain, indigestion, diarrhea and constipation. The GSRS has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms. The effect of the interventions on the GSRS will be assessed by a linear mixed model and will take into account information on this from all 7 days of treatment.
Change in Short Chain Fatty Acids (SCFA) in the stool | Throughout 14 days of product intake
  Measured using Gas Chromatography (GC)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Innovation Lab, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Siegwald L, Cherta-Murillo A, Christen S, Boulange CL, Chou CJ, Foata F, Lahiry A, Frezal A, Giner MP, Godin JP, Sakwinska O. The Impact of Low-Lactose, High Galacto-Oligosaccharides Milk on Gut Microbiome and Plasma Metabolome in Healthy Adults: A Randomized, Double-Blind, Controlled Clinical Trial Complemented by Ex Vivo Experiments. Curr Dev Nutr. 2025 Jul 24;9(9):107506. doi: 10.1016/j.cdnut.2025.107506. eCollection 2025 Sep. PMID 40909168